CLINICAL TRIAL: NCT01151462
Title: Postnatal HCMV Infection in Very Preterm Infants. Implications on Acute and Chronic Morbidity, Growth and Neurodevelopmental Outcomes Part of the Study on "Nutrition, Growth and Development Among Very Preterm Infants".
Brief Title: Postnatal HCMV Infection in Very Preterm Infants. Implications, Morbidity, Growth and Neurodevelopmental Outcomes.
Status: Withdrawn | Type: Observational
Why Stopped: The study was terminated prior to enrollment
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Ullevaal University Hospital (Other); University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Kenneth Strømmen, Arild Rønnestad, PhD, Oslo University Hospital
Other Study IDs: REK 2009/2249b
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2022-09-23 (Actual); Status verified 2013-05

CONDITIONS: Hearing Loss; Mental Retardation; Microcephaly; Chorioretinitis
Keywords: Postnatal HCMV infection in very preterm infants; Neurodevelopmental disabilities; Hearing loss; Mental retardation; Microcephaly; Chorioretinitis; Growth
MeSH Terms: conditions — Hearing Loss; Intellectual Disability; Microcephaly; Chorioretinitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum. Mothersmilk. Urine.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to investigate short and long term consequences from early postnatal HCMV infection transmitted via human milk in very preterm infants (birth weight < 1500 g or gestational age < 32 weeks). These infants are at high risk of early death or survival with chronic disease and neurodevelopmental impairment if infected with HCMV. Infection is a common complication in this group of patients and reported to be the most frequent cause of death after the second week of life. Systemic infection in the newborn period is reported as representing an independent risk factor for survival with neurodevelopmental impairment among very preterm infants.

DETAILED DESCRIPTION:
Approximately 70 % of fertile women in Norway are seropositive for HCMV. In practically all seropositive women a reactivation of the HCMV occurs during late pregnancy and lactation. In 75 - 80 % of HCMV seropositive lactating women this reactivation can be detected as presence of infectious HCMV in breast milk and witch is pathogenic and fully capable of causing infection in both term and preterm infants. Norway is one of few countries in the world where the provision of raw unpasteurized milk from the mothers to their very premature infants is encouraged regardless of the mothers HCMV status. Within the first few days after inclusion the mothers HCMV status will be established by serological tests. Weekly samples will be collected from the mother's breast milk and the baby's urine and frozen at minus 80 degrees Celsius for later quantitative analysis for the presence of HCMV virus by PCR technique. The plan is to enrol 260 very preterm infants over a period of 2 years. Exclusion criteria are congenital malformations, chromosomal abnormalities and clinical syndromes known to affect growth, and critical illness with short life expectancy. We wish to preform Magnetic Resonance Imaging (MRI) of the brain at term and 5 months corrected age. A parent-completed Questionnaire called the Ages and Stages Questionnaire (ASQ), will be sent to the infants' parents at 6, 12 and 20 months CA. We will perform a Visual Evoked Potential (VEP) test and an eye-tracking test at 5 months CA. During the 3rd year of life we will test children's ability to insert differently formed object into fitting apertures. The aim of this study is to investigate short and long term consequences from early postnatal HCMV infection transmitted via human milk in very preterm infants (birth weight < 1500 g or gestational age < 32 weeks). These infants are at high risk of early death or survival with chronic disease and neuro-developmental impairment if infected with HCMV. HCMV infection is a common complication in this group of patients and reported to be the most frequent cause of death after the second week of life. This study on postnatal HCMV infection will, together with the main study on nutrition (Nutrition, growth and development among very preterm infants, NCT01103219), provide results that will create a foundation for evidence based recommendations regarding optimal nutrition of very preterm infants. Much uncertainty is attached to the consequences from providing raw human milk from HCMV seropositive mothers to their very preterm infants. Raw HCMV positive human milk given to very preterm infants may lead to unwanted consequences on health on a scale that is largely unknown and may be underrated.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight below 1,500 grams
* Written parental consent
* Infants receiving their own mothers milk

Exclusion Criteria:

* Congenital malformations
* Critical illness with short life expectancy

Min Age: 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Premature infants with birth weight below 1,500 grams born at Oslo University Hospital and Akershus University Hospital.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Positive HCMV PCR in urine > 2 weeks after birth is diagnostic for postnatal HCMV infection. | > 2 weeks after birth

SECONDARY OUTCOMES:
Incidence and consequences of postnatal HCMV infection in terms of neurodevelopment disabilities including cognition, vision, hearing, movement and growth. | Before 5 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Arild Rønnestad, Dr.med (PhD), Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway

REFERENCES:
- [Background] Ronnestad A, Abrahamsen TG, Medbo S, Reigstad H, Lossius K, Kaaresen PI, Egeland T, Engelund IE, Irgens LM, Markestad T. Late-onset septicemia in a Norwegian national cohort of extremely premature infants receiving very early full human milk feeding. Pediatrics. 2005 Mar;115(3):e269-76. doi: 10.1542/peds.2004-1833. Epub 2005 Feb 1. PMID 15687416
- [Background] Ronnestad A, Abrahamsen TG, Medbo S, Reigstad H, Lossius K, Kaaresen PI, Engelund IE, Irgens LM, Markestad T. Septicemia in the first week of life in a Norwegian national cohort of extremely premature infants. Pediatrics. 2005 Mar;115(3):e262-8. doi: 10.1542/peds.2004-1834. Epub 2005 Feb 1. PMID 15687417
- [Background] Markestad T, Kaaresen PI, Ronnestad A, Reigstad H, Lossius K, Medbo S, Zanussi G, Engelund IE, Skjaerven R, Irgens LM; Norwegian Extreme Prematurity Study Group. Early death, morbidity, and need of treatment among extremely premature infants. Pediatrics. 2005 May;115(5):1289-98. doi: 10.1542/peds.2004-1482. PMID 15867037
- [Background] Henriksen C, Haugholt K, Lindgren M, Aurvag AK, Ronnestad A, Gronn M, Solberg R, Moen A, Nakstad B, Berge RK, Smith L, Iversen PO, Drevon CA. Improved cognitive development among preterm infants attributable to early supplementation of human milk with docosahexaenoic acid and arachidonic acid. Pediatrics. 2008 Jun;121(6):1137-45. doi: 10.1542/peds.2007-1511. PMID 18519483
- [Background] Westerberg AC, Henriksen C, Ellingvag A, Veierod MB, Juliusson PB, Nakstad B, Aurvag AK, Ronnestad A, Gronn M, Iversen PO, Drevon CA. First year growth among very low birth weight infants. Acta Paediatr. 2010 Apr;99(4):556-62. doi: 10.1111/j.1651-2227.2009.01667.x. Epub 2010 Jan 20. PMID 20096031